CLINICAL TRIAL: NCT00194766
Title: Continuous Temozolomide (SCH 52365) in Patients With Advanced or Metastatic Soft Tissue Sarcoma or Metastatic Breast Cancer, Phase II
Brief Title: Continuous Temozolomide in Patients With Advanced or Metastatic Soft Tissue Sarcoma or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Schering-Plough (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-1283-A
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer; Soft Tissue Sarcoma
Keywords: Breast cancer; Soft tissue sarcoma
MeSH Terms: conditions — Breast Neoplasms; Sarcoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Temozolomide 75 mg/m2 daily for 6 weeks followed by a two week rest period for a total cycle length of 8 weeks. Treatment is repeated until disease progression, excessive toxicity or other reason to suspend protocol treatment.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide 75 mg/m2 daily for 6 weeks followed by a two week rest period for a total cycle length of 8 weeks. Treatment is repeated until disease progression, excessive toxicity or other reason to suspend protocol treatment.

SUMMARY:
The purpose of this study is to determine whether treatment with temozolomide can effect the survival of patients with advanced breast cancer or soft tissue sarcoma.

DETAILED DESCRIPTION:
Because repeated dosing of temozolomide correlates with an improved response, which may be due to progressive depletion of the enzyme AT, our hope is that a daily oral schedule will be the most active schedule of this agent. In phase I studies doses below 85 mg/m2/day continuously have been well-tolerated. We plan to begin dosing at 75 mg/m2/day for 6 weeks out of an 8 week cycle and to escalate to 85 and 100 mg/m2/day in patients who have no grade 3/4 toxicity.

The purpose of this study is to determine whether treatment with temozolomide can effect the survival of patients with advanced breast cancer or soft tissue sarcoma. To do this we will assess the response rate, time to progression, and survival in patients with advanced breast cancer or soft tissue sarcoma who are treated with temozolomide.

ELIGIBILITY:
Inclusion Criteria:

Patients must have either:

* Stage IV, microscopically-confirmed carcinoma of the breast with:

  * Relapse or progression while receiving, or within 12 months of having received, an anthracycline-containing (doxorubicin or mitoxantrone) or taxane-containing (paclitaxel or docetaxel) regimen as either adjuvant treatment or therapy for advanced breast cancer, or
  * Treatment to a maximum dose of anthracycline (e.g., greater than 450 mg/m2 of doxorubicin), or
  * A dose-limiting toxicity from a taxane, or
  * An ECOG performance status of 2.

    * OR -
* Unresectable or metastatic, microscopically-confirmed soft tissue sarcoma, that is not amenable to treatment with Adriamycin or Ifosfamide due to:

  * Poor cardiac reserve, or
  * Poor performance status (ECOG performance status = 2) or
  * Having failed treatment with Adriamycin or reached dose-limiting toxicity from chemotherapy.

Patients must have histologic slides and/or blocks must be available for review.

Patients must have measurable (bidimensionally) or evaluable disease.

Patients must be 18 years old or older.

Patients must have Karnofsky Performance Status greater than 70% (ECOG less than 2) at screen and on the first day of treatment.

Patients must have a life expectancy more than 16 weeks.

Patients must be informed consent must be obtained prior to enrollment.

Patients must be more than 2 weeks from prior surgery; more than 3 weeks from radiation therapy to the pelvis, spine or long bones; more than 3 weeks from prior chemotherapy (more than 6 weeks for mitomycin C or nitrosureas), or more than 2 weeks from prior hormonal therapy.

Exclusion Criteria:

Granulocytes less than 1,500/mm3.

Platelet count less than 100,000/mm3.

Hemoglobin less than 10 gm/dl.

Creatinine greater than 2.0 mg/dl.

Total bilirubin greater than ULN (institutional upper limit of normal).

Visceral crisis characterized by rapidly progressive hepatic or lymphangitic lung metastases (i.e. patients whose disease is beyond control).

Medically unstable (i.e. with uncontrolled disease); diagnosis of other systemic cancer.

Pregnancy or lactation; failure to employ adequate contraception.

Uncontrolled CNS disease.

Greater than 30% marrow previously irradiated.

Psychological, familial, sociological or geographical conditions which do not permit weekly medical follow-up and compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Response rate | <= 78 months

SECONDARY OUTCOMES:
Time to disease progression | <= 78 months
Survival | <= 78 months
To determine the toxicity of the regimen. | <= 78 months

CONTACTS AND LOCATIONS:
Overall Officials: James Butrynski, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington/Seattle Cancer Care Alliance, Seattle, Washington, United States